CLINICAL TRIAL: NCT01445964
Title: An Open-label, Single-dose, Three-treatment, Three-period Study to Investigate the Effect of SLCO2B1 Genotype and Apple Juice on Pharmacokinetics of Atenolol After Oral Administration in Healthy Male Korean
Brief Title: Effect of SLCO2B1 Genotype and Apple Juice on Pharmacokinetics of Atenolol After Oral Administration in Healthy Male Korean
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, In-Jin Jang, MD, PhD, Professor of Clinical Pharmacology and Therapeutics, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUCPT11_ATE; Pan Asian-Atenolol-1
Record Dates: First submitted 2011-04-29; First posted 2011-10-04 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: SLCO2B1 genotype; effect of apple juice
MeSH Terms: interventions — Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): SLCO2B1 wild type allele
  Interventions: Drug: Atenolol; Drug: Atenolol with apple juice 1200 mL; Drug: Atenolol with apple juice 600 mL
- 2 (Experimental): SLCO2B1 variant allele
  Interventions: Drug: Atenolol; Drug: Atenolol with apple juice 1200 mL; Drug: Atenolol with apple juice 600 mL

INTERVENTIONS:
Drug: Atenolol — Atenolol oral administration
Drug: Atenolol with apple juice 1200 mL — Atenolol oral administration with apple juice 1200 mL
Drug: Atenolol with apple juice 600 mL — Atenolol oral administration with apple juice 600 mL

SUMMARY:
An open-label, single-dose, three-treatment, three-period study to investigate the effect of SLCO2B1 genotype and apple juice on pharmacokinetics of atenolol after oral administration in healthy male Korean.

ELIGIBILITY:
Inclusion Criteria:

* Subject is informed of the investigational nature of this study and voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB) - approved informed consent prior to performing any of the screening procedures

Exclusion Criteria:

* A subject with history of allergies including study drug (atenolol) or other drug allergies (aspirin, antibiotics, etc.), or history of clinically significant allergies

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
AUC of atenolol according to the SLCO2B1 genotypes | 0-48 hr after drug administration
  The area under the plasma concentration versus time curve, from time 0 to the last measurable concentration, as calculated by the linear/log trapezoidal method will be summarized by treatment and genotype group using descriptive statistics.

SECONDARY OUTCOMES:
Blood pressure of the subjects who administered atenolol according to the SLCO2B1 genotypes | 0-48 hr after drug admnistration
  Blood pressure measurement will be presented as descriptive statistics for the difference from baseline where appropriate.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 0-48 hr after drug admnistration
  Number of participants with adverse event as a measure of safety and tolerability
  *Measure of safety and tolerability: physical examinations, ECG, Laboratory tests (including hematology, chemistry, urinalysis)
  - Descriptive statistics will be calculated for quantitative safety data as well as for the difference from baseline where appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea